CLINICAL TRIAL: NCT04987385
Title: Effect of Protein Supplementation on Plasma Sodium Levels and Urinary Urea Excretion in Patients With SIAD - a Monocentric Open- Label Proof-of-concept Study -The TREASURE Study
Brief Title: Effect of Protein Supplementation on Plasma Sodium Levels and Urinary Urea Excretion in Patients With SIAD
Acronym: TREASURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01116; kt21ChristCrain2
Record Dates: First submitted 2021-07-21; First posted 2021-08-03 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Syndrome of Inappropriate Antidiuresis (SIAD)
Keywords: protein supplementation; plasma sodium level; hyponatremia; urea
MeSH Terms: conditions — Inappropriate ADH Syndrome; Hyponatremia | interventions — Urea

STUDY DESIGN:
Intervention Model Description: proof-of-concept study, no control group needed since patients serve as their own control in the second treatment phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm: Phase 1: protein supplementation, Phase 2: Urea (Other)
  Interventions: Dietary Supplement: Protein supplementation; Dietary Supplement: Oral urea

INTERVENTIONS:
Dietary Supplement: Protein supplementation — Patients will receive a box with 7 sealable of 90-gram protein containers that will be dissolved in maximal 1L liquid (i.e., water or milk) that should be integrated in the usual daily hydration volume documented at baseline and taken daily for the following 7 days, while keeping their usual meal composition and usual fluid intake. A wash-out period of minimum 7 days between Protein supplementation and Oral urea will be performed.
Dietary Supplement: Oral urea — Patients will receive a box with 7 30-grams urea sealable containers. The total daily oral urea dosage of 30 grams that will be dissolved in maximal 1L of a liquid of choice (water, milk, juice, …) that should be integrated in the usual daily hydration volume documented at baseline and taken daily for the following 7 days, while keeping their usual meal composition and usual fluid intake.

SUMMARY:
This study aims to investigate whether a 7-day dietary high protein supplementation of 90 grams per day increases plasma sodium levels in hyponatremic patients with chronic SIAD.

Enrolled patients will receive first dietary high protein supplementation for one week. After a wash-out phase of at least one week, the patients will receive oral urea for another week.

DETAILED DESCRIPTION:
Hyponatremia (blood sodium <135 mmol/l) is the most frequent electrolyte and fluid disturbance with a prevalence up to 30% in hospitalized patients. The most common etiology of euvolemic hyponatremia is the syndrome of inappropriate antidiuresis (SIAD) which is also the main etiology of hyponatremia overall. Urea osmotic diuresis has been reported to cause hypernatremia in critically ill patients in intensive care unit (ICU), showing that urea can influence sodium levels. Increasing solute intake with oral urea represents a valid treatment approach to increase urine volume and solute free water clearance through osmotic diuresis and reduction of urinary sodium excretion in SIAD. In Switzerland, urea is a medical food prepared as a compounding agent by pharmacies. Endogenous proteins and dietary protein are metabolized into nitrogen which is metabolized to soluble excretable urea by the liver. Protein intake could represent an osmotic relevant source of urea. The Jone's factor of 6,25 is commonly used to convert nitrogen to protein equivalent, assuming an average nitrogen content of 16% in protein (100g protein / 6,5 = 16g nitrogen).

Urea (CH₄N₂O) contains 46,6% nitrogen (atomic weight of nitrogen = 14 g/mol, atomic weight of urea = 60,1 g/mol). Using these ratios, 30g urea would correspond to 14g nitrogen and 87,5g protein. In this study, a 90g protein supplementation will be used, which corresponds roughly to 30g urea, in form of a daily intake of protein powder (Whey Protein®, foodspring GmbH, Germany or Clear Whey Isolate®, MyProtein THG Company, United Kingdom), which is freely marketed as food in Switzerland. Both interventional products are not considered as drugs.

Patients with a plasma sodium concentration <125 mmol/L are at increased risk for overcorrection, i.e., an increase in plasma sodium levels >10 mmol/L in the first 24 hours of treatment. An additional visit will be planned on the second day of treatment in order to recognize rise over this limit and initiate relowering counteractions, which will include the skip of the second powder intake and oral fluid intake.

This study is to analyze whether protein supplementation can increase plasma sodium levels in patients with SIAD by increasing urinary urea excretion.

ELIGIBILITY:
Inclusion Criteria:

* previous documented diagnosis of chronic SIAD
* confirmed diagnosis of SIAD at screening visit defined as:

  * plasma sodium concentration <135 mmol/L, measured in lithium heparin plasma
  * Plasma osmolality <300 mOsm/kg
  * Urine osmolality >100 mOsm/kg
  * Urine sodium concentration >30mmol/l
  * Clinical euvolemia, defined as an absence of signs of hypovolemia (orthostasis, tachycardia, decreased skin turgor, dry mucous membranes) or hypervolemia (edema, ascites)

Exclusion Criteria:

* lactose intolerance, celiac disease, milk protein allergy, soja allergy, nuts allergy or known hypersensitivity or allergy to one of the components of the protein supplementation (Whey Protein®, foodspring GmbH, Germany or Clear Whey Isolate®, MyProtein THG Company, United Kingdom)
* inborn metabolic disorders implying carbohydrate, lipid or protein metabolism - severe symptomatic hyponatremia in need of treatment with 3% NaCl-solution or in need of intensive/intermediate care treatment at time of inclusion
* Risk factors for osmotic demyelination syndrome: hypokalaemia (K <3,4 mmol/L), malnutrition, advanced liver disease, alcoholism.
* contraindication for lowering blood pressure
* type 1 diabetes mellitus
* uncontrolled type 2 diabetes mellitus (defined as HbA1c >8.0%)
* uncontrolled hypothyroidism
* uncontrolled adrenal insufficiency
* reduction of eGFR <60 mL/min/1,73 m2 (KDIGO G3, G4 and G5) or end stage renal disease (dialysis)
* severe hepatic impairment (ALAT/ASAT >3x upper limit) or advanced symptomatic liver disease defined as past or current hepatic encephalopathy, liver cirrhosis Child C or decompensated (bleeding, jaundice, hepatorenal syndrome).
* treatment with a diuretic, a SGLT2 inhibitor or a corresponding combined preparation, lithium chloride, urea, vaptans, demeclocycline in the two weeks before screening.
* severe immunosuppression defined as leucocytes <2G
* pregnancy, wish to become pregnant during study period or breastfeeding
* end of life care
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Current participation in another intervention study
* lack of capacity or other reason preventing from giving informed consent or following study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Change in plasma sodium concentration, (mmol/l) | from baseline to 7 days after protein supplementation (7 days)
  The change of blood sodium during protein supplementation regimen will be visualized by means of line plots and boxplots for patients with chronic SIAD.

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR), (ml/min/1,73m2) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in estimated glomerular filtration rate (eGFR)
Change in blood and urine osmolality, (mOsm/kg) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in blood and urine osmolality
Change in blood and urine potassium, (mmol/L) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in blood and urine potassium
Change in blood and urine creatinine, (umol/L) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in blood and urine creatinine
Change in blood and urine urea, (mmol/L) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in blood and urine urea,
Change in blood and urine uric acid, (umol/L) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in blood and urine uric acid
Change in blood and urine glucose, (mmol/L) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in blood and urine glucose
Change in copeptin, (pmol/l) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in copeptin
Change in aldosterone, (pmol/l) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in aldosterone
Change in renin, (mIU/L) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in renin
Change in MR-proANP, (pmol/l) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in MR-proANP
Change in NT-proBNP, (pmol/L) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in NT-proBNP
Change in oral daily fluid intake, (ml) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in oral daily fluid intake assessed by a self-completed drinking protocol
Change in body weight, (kg) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in body weight (kg)
Change in both systolic and diastolic blood pressure, (mmHg) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in both systolic and diastolic blood pressure (mmHg)
Change in heart rate, (beats/minute) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in heart rate (beats/minute)
Change in general well-being measured by visual analogue scale (VAS, 0-10) | from baseline to 7 days after urea supplementation (up to 21 days)
  Change in general well-being measured by visual analogue scale (VAS, 0-10), with a range from 0 "worst well-being" to 10 "excellent well-being".
Number of signs of hyponatremia (vertigo, headache, nausea, attention deficit, mental slowness, forgetfulness, gait instability) assessed by a questionnaire (yes/no) | from baseline to 7 days after urea supplementation (up to 21 days)
  number of signs of hyponatremia (vertigo, headache, nausea, attention deficit, mental slowness, forgetfulness, gait instability) assessed by a questionnaire (yes/no)
Short-term change in plasma sodium level (mmol/L) | at day 1 (after treatment start)
  Short-term change in plasma sodium levels in patients with a plasma sodium concentration <125 mmol/L at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. med., Principal Investigator — Universitätsspital Basel, Endokrinologie, Diabetologie und Metabolismus
Locations (1):
- University Hospital Basel, Department of Endocrinology, Basel, Switzerland